CLINICAL TRIAL: NCT04507191
Title: Prognostic Value of PDL1 in Ovarian High Grade Serous Carcinoma
Brief Title: PDL1 in Ovarian High Grade Serous Carcinoma
Status: Completed | Type: Observational
Sponsor: Port Said University hospital (Other)
Collaborators: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mayada saad, Lecturer of pathology, Port Said University hospital
Other Study IDs: R.20.07.957
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: immunohistochemical staining — immunohistochemical staining of programmed death-ligand 1 (PDL1) marker

SUMMARY:
the main purpose is to study the prognostic effect of PDL1 in ovarian cancer especially HGSC. Therefore, in the present study the investigators analyzed the expression of PDL1in HGSC by immunohistochemistry, and results were correlated to prognosis.

DETAILED DESCRIPTION:
this cross-sectional study on 54 specimens of primary ovarian high grade serous carcinoma cases who attended to Oncology Centre, Mansoura University, Mansoura, Egypt in the period from 2012 till 2019. The cases were chosen randomly. All clinicopathological data including tumor stage (T), L.N metastases (N), metastasis (M), (FIGO) staging system, ascites, recurrence, residual tumor, CEA level, CA125 level, and peritoneal deposits analyzed. The investigator followed the clinical outcomes in the form of disease free survival (DFS) and overall survival (OS). The mean duration of follow up will be 43.4 months. The OS were calculated from the time of diagnosis to death. DFS is the time from the end of therapy to first recurrence or metastases. the specimens were stained with PDL1 marker in pathology department Port Said university.

Statistical analysis: Data was analyzed using SPSS software V.16. Continuous data was presented in the form of mean (SD) or Median (min-max) according to the results of Shapiro-Wilk testing for the assumptions of normal distributions of data. Categorical data will be presented in the form of frequencies and percentages. Statistical significance will be tested by Welch's t-test, or Mann-Whitney U for continuous data (with respect to presence or absence of normal distribution of data). Also, chi square test or Fisher's Exact Test will be performed for categorical data (with respect to the minimal expected values in the contingencies tables). Correlations of different tumour markers will be calculated using Spearman's rho Coefficient. Kaplan-Meier test was used to test for overall survival and disease free survival of patients with respect to tumour expression of PDL1. Comparisons will be done using Log Rank (Mantel-Cox). Significance level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with primary ovarian cancer

Exclusion Criteria:

* patients with metastatic ovarian cancer

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients diagnosed with primary serous ovarian cancer and subjected to staging laparotomy
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
number of slides stained positive to PDL1 marker | 7 years from 2012 to 2019
  using immunohistochemical staining for PDL1 markers for all slides of cases with ovarian tumor

SECONDARY OUTCOMES:
correlation between PDL1 expression to clinicopathological parameters of ovarian high grade serous carcinoma | 7 years from 2012 to 2019
  correlation between PDL1 expression to criteria as ascites, peritoneal nodules and metastasis

OTHER OUTCOMES:
correlation between PDL1 expression to prognosis of ovarian high grade serous carcinoma | 43.3 months
  correlation between PDL1 expression to cancer free peroid

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Port Said University, Port Said, Egypt

IPD SHARING:
Plan to Share IPD: Undecided